CLINICAL TRIAL: NCT05513105
Title: Iron Study of Neonates: Factors Affecting and Impact on Their Health Status at Birth in Assuit University Children's Hospital
Brief Title: Iron Study of Neonates Iron Study of Neonates Birth in Assuit University Children's Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Hashem, Principle investigator, Assiut University
Other Study IDs: Asiout
Record Dates: First submitted 2022-08-21; First posted 2022-08-24 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Iron Study of Neonates: Factors Affecting and Impact on Their Health Status at Birth in Assuit University Children's Hospital

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Iron study of neonates — Blood sambles

SUMMARY:
Iron study of neonates: factors affecting and impact on their health status at birth in Assuit University Children's Hospital

DETAILED DESCRIPTION:
Iron is an essential micronutrient that plays a significant role in critical cellular functions in all organ systems in all species. Iron is particularly vital for early brain growth and function in humans since it supports neuronal and glial energy metabolism, neurotransmitter synthesis and myelination [1-5]. The need to establish standard curves for cord serum ferritin concentrations throughout the third trimester of pregnancy is based on the risk of developing brain iron deficiency as storage iron pools become depleted in certain gestational conditions [6-8]. Iron deficiency during the fetal or postnatal periods can alter brain structure, neurochemistry and cognitive functioning, and lead to long-term cognitive and motor impairment that cannot be corrected by iron supplementation [9-11]. Newborn infants with the lowest quartile of cord ferritin concentrations (<76 μg/l) have impaired mental and psychomotor function at school age [12]. Iron-deficient infants of diabetic mothers (IDM) with low neonatal ferritin concentrations (<35 μg/l) have impaired auditory recognition memory processing at birth compared with iron-sufficient IDM (ferritin >35 μg/l) [13]. Pre-term infants with low serum ferritin concentrations (<75 μg/l) at 37 weeks post-conception have abnormal neurologic reflexes [14].

Direct measurement of brain iron in newborn infants is not currently feasible.Total body iron and iron storage estimates are based on measurements of serum markers, such as hemoglobin (Hgb) and ferritin concentrations [15]. Serumferritin concentration has been used as a standard measurement of iron stores ininfants, children and adults [16-19]. The relationships between ferritin concentrations and total body storage iron in these populations are well established. In adults, 1 μg/l of serum ferritin is equivalent to 8-10 mg ofstorage iron [20]. In newborn infants, the ratio of serum ferritin to liver nonheme iron concentration is closer to 1:2.7 [21]. In spite of the wide availability of serum ferritin as a screening test, normative data at birth, as a function of specific gestational ages from 23 to 41 weeks,

Low serum ferritin concentrations are seen only in iron deficiency. Elevated ferritin concentrations in the newborn can be a consequence of neonatal hemochromatosis, excessiveiron administration or RBC transfusions. Serum ferritin concentrations are also elevated during periods of infection,inflammation and neoplasia. Under these conditions, serum ferritin behaves as an acute-phase reactant that can mask the diagnosis of iron deficiency [22]. Iron requirements in women are significantly higher in the pregnant state than in the nonpregnant state. The total iron requirement of a full-term pregnancy is approximately 1,000 mg [23]. Iron requirements for pregnant women increase significantly in the second and third trimesters, with the expansion of maternal blood volume and fetal red cell mass [23]. The fetus accumulates iron at a rate of 1.35 mg/kg of fetal weight in the third trimester, maintaining an average iron content of 75 mg/kg of body weight during the last trimester [24.25]. At term, 70-80% of fetal iron is present in RBCs as Hgb, 10% in tissues as myoglobin and cytochromes, and the remaining 10-15% stored in reticuloendothelial and parenchymal tissues as ferritin and hemosiderin [24]. The placenta serves as the regulatable conduit for maternal-fetal iron transport. The amount of iron passing through the placenta increases with gestation. Iron is transferred against a concentration gradient from the placenta to the fetus, especially during the later stages of pregnancy. The placenta can also serve as a storage organ for iron during pregnancy.

Factors that influence neonatal ferritin concentration at birth include duration of gestation, fetal sex, maternal iron status and conditions altering maternal-fetal iron exchange.. At- or near-term female newborn infants have higher cord serum ferritin concentrations than male

ELIGIBILITY:
Inclusion Criteria:

* Neonates delivered at women Assuit university hospital either ceserian or normal vaginal delivery

Exclusion Criteria:

* *Congenital malformation

  * history of genetics or chromosomal disease
  * history of inborn errors of metabolic disease
  * Neonates who we cannot catch cord blood sample immediate afer birth

Ages: 1 Minute to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: NeonateS birth in Assuit University Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-19 (Estimated); Primary Completion 2023-01-12 (Estimated); Study Completion 2023-12-22 (Estimated)

PRIMARY OUTCOMES:
Iron study of neonates | 3years
  describes iron study of neonates affecting health status at birth

IPD SHARING:
Plan to Share IPD: Undecided